CLINICAL TRIAL: NCT02579408
Title: Controlled Attenuation Parameter for the Evaluation of Donor Steatosis in Living Donor Liver Transplantation
Brief Title: Quantifying Steatosis in Liver Transplant Donors
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wai-Kay Seto, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: CAP LDLT
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Non-alcoholic Fatty Liver Disease; Evidence of Liver Transplantation
Keywords: NAFLD; LDLT; steatosis; CAP; transient elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma for storage in anticipation of future biomarkers for the prediction of improved post-transplant outcomes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LDLT donor: Donors of living donor-related liver transplantation

SUMMARY:
Non-alcoholic fatty liver disease is the most common chronic liver disease in Hong Kong. Its presence among donors of living donor liver transplants could affect the outcomes of recipients of liver transplantation. By using controlled attenuation parameter (CAP) measurements, the investigators aim to investigate the association of CAP measurements and severity of fatty liver among liver donors in the recipient outcomes of living donor liver transplantation.

DETAILED DESCRIPTION:
Living donor liver transplantation (LDLT) has been increasing worldwide due to the critical shortage of cadaveric donors and the rising number of patients awaiting liver transplantation. The long-term survival rates of LDLT are now comparable to that of deceased donor liver transplantation. Currently, two-thirds of all liver transplants performed in Hong Kong are LDLT.

The ultimate goal of LDLT is to guarantee donor safety while optimizing the best possible recipient outcome. Donor liver steatosis is a well-known factor which could influence graft function and long-term outcomes of the recipient allograft, and also affects donor hepatic recovery. When needed, pre-operative liver biopsy is often used for the quantitative assessment of donor steatosis, with LDLT not recommended when steatosis exceeds 30%. Nonetheless, liver biopsy is limited by its invasive nature, sampling error and intra-observer variations. Imaging evaluation for the quantification of steatosis via ultrasonography or computed tomography also has various pitfalls. There is currently no universal consensus on the ideal method in assessing donor steatosis.

Controlled attenuation parameter (CAP) is a novel non-invasive method to quantify hepatic steatosis using ultrasonic attenuations to postulate fat content. It has been demonstrated to have good correlation with the degree of hepatic steatosis in both Western and Asian populations. The investigators aim to evaluate the application of CAP in the donor workup of LDLT and to investigate for its association with post-transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 LDLT donor who has completed donor workup
* Consents to study entry

Exclusion Criteria:

* Concomitant liver disease, including chronic hepatitis B and C infection, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson disease, and increased alcohol intake (30g per week for male, 20g per week for female).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Donors of living donor liver transplantation conducted in Queen Mary Hospital, Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recipient allograft short-term outcomes | Up to 30 days
  Includes:
  1. Intraoperative parameters (blood transfusion, operation time etc)
  2. Postoperative outcomes (ICU stay, hospital stay, hospital mortality, major postoperative complication etc) Initial poor function, defined as an AST or ALT >1,500 U/L on two consecutive measurements within the first 72 hours Primary graft nonfunction, defined as poor function of allograft culminating in either death of recipient or retransplant
Recipient allograft long-term outcomes | Up to 1 year
  Includes:
  1. Overall survival
  2. Primary graft nonfunction up to 1 year
  3. Liver stiffness measurements via transient elastography at 1 year
  4. Controlled attenuation parameter measurements at 1 year

SECONDARY OUTCOMES:
Association of controlled attenuation parameter scores with clinical parameters of LDLT donor | At time of transplant
  Correlation of controlled attenuation parameter measurements with:
  1. Body mass index (in kg/m2)
  2. Waist circumference (in cm)
  3. Liver volumetry and fat quantification via pre-operative computed tomography. Fat quantification is calculated by the hepatic attenuation measurement
  4. Donor histological grading of steatosis

CONTACTS AND LOCATIONS:
Overall Officials: Wai Kay Seto, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine and Department of Surgery, The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong